CLINICAL TRIAL: NCT01906437
Title: Non-invasive Detection of Cardiac Fibrosis After Administration of Doxorubicin-based Chemotherapy in Patients With Lymphoma Using Cardiac Magnetic Resonance
Brief Title: Cardiac Fibrosis by CMR in Patients With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tomas Neilan, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 11-443; NCT02055040 (obsolete NCT alias)
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Lymphoma
Keywords: Cardiac fibrosis and Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Magnetic Resonance: Cardiac Magnetic Resonance scan at visits 1 and 2
  Interventions: Device: Cardiac Magnetic Resonance Scan

INTERVENTIONS:
Device: Cardiac Magnetic Resonance Scan — Cardiac Magnetic Resonance Scan

SUMMARY:
A study to test the effectiveness of an investigational imaging technique for detecting cardiac injury after the administration of certain chemotherapies, such as doxorubicin. "Investigational" means that the imaging technique is still being studied and that research doctors are trying to find out more about it- such as whether the technique can detect lower levels of cardiac injury after treatment with doxorubicin. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved the use of gadolinium or approved the use of CMR studies for detection of cardiac toxicity after doxorubicin.

The chemotherapy drug that you have been scheduled to be treated with, doxorubicin, has been associated with the development of heart failure in some patients. Cardiac Magnetic Resonance (CMR) is a type of MRI scan that uses a magnetic field to produce pictures of the heart. The CMR scan has been used in other studies and information from those other research studies suggest that this imaging technique may help to better detect differences in the structure of the heart muscle after treatment with doxorubicin. In this research study, we hope that we can better detect changes in the heart muscle after treatment with doxorubicin with a CMR scan in the hopes that cardiac injury can be detected and treated earlier to ultimately prevent the possible development of heart failure

DETAILED DESCRIPTION:
If you choose to take part in this study, we will ask you to sign this consent form before we do any study procedures. All participants will come in for a CMR scan prior to their first treatment with doxorubicin

- Visit 1 Visit 1 will take place prior to starting chemotherapy. The visit will take about 1.5 hours. We will ask you to come to the Shapiro Cardiovascular Center at the Brigham and Women's Hospital or Massachusetts General Hospital for your study visit.

For subjects that qualify, we will bring you for the heart CMR scan, an echocardiogram and some blood work.

Blood testing: Before your CMR scan we will take some blood via the IV cannula. We will take about 4 tubes of blood. This is equivalent to 2 ½ tablespoons of blood. From this blood we will test for blood markers of cardiac injury and compare these results to your other tests.

CMR Scan: For the CMR scan, you will be asked to lie still on the scanner table that slides into a tunnel-shaped machine. Four electrocardiogram (EKG) patches with wires attached will be placed on your chest or your back to check your heart rate. We will place an intravenous (IV) catheter in one of your arms. An IV catheter is a thin plastic tube that is put into a vein with a needle. The IV catheter will be used to give you a CMR contrast dye (gadolinium). The dye will help us to identify subtle changes within the heart muscle. This dye, gadolinium, is used routinely in CMR studies. We will also draw a sample of blood from the IV catheter to measure your red blood cell count. Then, the scanner table will move slowly into the tunnel-shaped CMR machine so the pictures can be taken. The machine is slightly wider than your body and there may be little room to move. If you feel any discomfort or need to stop the test, you will be able to tell this to the research staff. You will be able to speak to them while you are having the CMR and they will be able to speak to you. If you think that you might be too anxious about being inside the narrow CMR scanner for a long period of time, we may prescribe a drug called to help relax you if you think it might be helpful.

The CMR scan will take one hour.

Echocardiogram: An echocardiogram is a test used by doctors to monitor heart function. An echocardiogram is a safe test that uses ultrasound to image the heart. After completion of the CMR test, you will have an echocardiogram. This test will take place in the same area as the CMR test. The echocardiogram test will take 40 minutes.

- Visit 2: Visit 2 will take place about 2-4 weeks after your last cycle of doxorubicin chemotherapy.

When you come back for Visit 2, you will have the same type of CMR scan, echocardiogram and blood testing that you had during Visit 1.

- Visit 3: At visit three we will perform an exercise test on a bicycle. The test is designed to test the oxygen consumption of your body when exercising. It provides a way of quantifying the ability of the body to exercise. This test will take 30 minutes. During this test subjects sit on the bicycle for at least 3 minutes pedaling at a rate of 60 cycles per minute and slowly the work-load is increased until peak exercise is obtained. We define peak exercise as being tired or breathless. Heart rate and blood pressure are recorded during the test. During the test you will breathe through a mouthpiece from which we will measure oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 and able to give consent
* New diagnosis of lymphoma and scheduled to undergo doxorubicin (DOX)-based chemotherapy.

Exclusion Criteria:

* Concurrent radiotherapy prior to the performance of both CMR studies, however consolidative radiotherapy after the completion of DOX and after the acquisition of the second CMR study is acceptable
* No prior malignancy treated with chemotherapy or mediastinal radiotherapy
* No contraindications to the performance of a magnetic resonance study:
* The presence of an implanted metallic object such as a cardiac pacemaker or implantable defibrillator
* An implanted neural stimulator
* Any ferromagnetic implants not deemed MRI-safe
* Intra-ocular metallic foreign bodies
* Severe claustrophobia
* Pregnancy
* Inability to perform an exercise test
* Glomerular filtration rate < 60 ml/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Myocardial ECV | 2 Years
  - To determine if a novel cardiac magnetic resonance-based index, the extracellular volume fraction (ECV), of myocardial fibrosis is altered early after doxorubicin-based chemotherapy.

SECONDARY OUTCOMES:
Alteration of serum biomarkers after doxorubicin based chemotherapy | 2 years
  - To determine if serum biomarkers of cardiac stress, collagen turn-over, and myocardial injury are altered after doxorubicin-based chemotherapy
Alteration of echocardiographic indices after doxorubicin-based chemotherapy | 2 Years
  - To determine if conventional and novel echocardiographic indices are altered after doxorubicin-based chemotherapy.
Measurement of cardiopulmonary functional capacity | 2 years
  - To determine if measures of cardiopulmonary functional capacity are abnormal after doxorubicin-based chemotherapy.
Determine association between measurements pre- and post-doxorubicin-based chemotherapy | 2 Years
  - To determine if there is an association between CMR, echocardiographic, serum, and functional measures pre- and post doxorubicin-based chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Neilan, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Insitute, Boston, Massachusetts